CLINICAL TRIAL: NCT06178926
Title: Efficacy and Safety of Ciprofol Sedation in Patients Undergoing Liver Cancer Percutaneous Radiofrequency Ablation: A Double-Blind, Randomized, Noninferiority Trial
Brief Title: Ciprofol Sedation in Patients Undergoing Liver Cancer Percutaneous Radiofrequency Ablation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Wang Jiangling, Principle Investigator, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-2023-350
Record Dates: First submitted 2023-07-25; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Liver Cancer; Ciprofol
Keywords: Radiofreqency ablation; Liver Cancer; Ciprofol
MeSH Terms: conditions — Liver Neoplasms | interventions — Propofol; (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol; HSK3486

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol (Active Comparator): Use propofol for sedation during anesthesia.
  Interventions: Drug: Propofol
- Ciprofol (Experimental): Use ciprofol for sedation during anesthesia
  Interventions: Drug: Ciprofol

INTERVENTIONS:
Drug: Propofol — Propofol was IV infused 1.0-1.5mg/Kg and then maintenance at 1.0-2.0mg/Kg/h
  Other Names: Diprivan; Propoven
  Arms: Propofol
Drug: Ciprofol — Ciprofol was IV infused 0.2- 0.3mg/Kg and then maintenance at 0.2-0.3mg/Kg/h
  Other Names: HSK3486
  Arms: Ciprofol

SUMMARY:
Efficacy and Safety of Ciprofol Sedation in Patients Undergoing Liver Cancer Percutaneous Radiofrequency Ablation

DETAILED DESCRIPTION:
Ciprofol was injected before ablation and sedation scores were measured to make sure certain sedation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who intend to undergoing ultrasound-guided percutaneous radiofrequency ablation of liver tumors;
* Age: 18-75 years old;
* ASA grade I-III;
* Laboratory examination meets the following conditions: neutrophils >1.5×109/L, platelet >80×109/L, hemoglobin >90g/L, aspartate transferase <1.5×ULN, total bilirubin <1.5×ULN, serum creatinine <1.2 x ULN;
* Chemotherapy < 4 times.

Exclusion Criteria:

* Patients who are known to be allergic to propofol, opioids, eggs, soy products, or patients who are contraindicated with these drugs or foods due to illness;
* serious organ dysfunction and other systemic diseases, such as liver dysfunction, renal dysfunction; Worsening congestive heart failure within the last 6 months resulting in hospitalization or adjustment of medication; Severe aortic or mitral stenosis; Heart surgery (heart valve replacement) within the last 6 months; Acute myocardial infarction in the last 6 months; Hemodynamic disturbance due to arrhythmia; Respiratory diseases; Cerebrovascular diseases; . Taking propofol, opioids or other analgesic and sedative drugs 72 hours before . Emergency surgery;
* Those who are unable to communicate with the researcher normally or who are deemed unsuitable by the researcher and refuse to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Sedation efficacy | From the start of propofol/ciprofol injection to 4 min after sedation.
  Satisfaction assessed by MOAAS, Modified Observer's Assessment of Alertness and Sedation (MOAA/S) scale is a validated 6-point scale assessing responsiveness of patients coinciding with the American Society of Anesthesiologists (ASA) continuum of sedation. MOAA/S 0 to 1 represent deeper sedation, MOAA/S 2 to 3 represent moderate sedation and MOAA/S 4 to 5 represent lighter to no sedation. In this study, MOAAS between 2-3 after initial IV dosage of propofol/ciprofol was defined as efficacy sedation.

SECONDARY OUTCOMES:
Respiratory depression | From the injection of propofol/ciprofol to the period patient return to the ward, an average of 2 hours.
  Any respiratory depression from the injection of propofol/ciprofol to fully recovery after surgery. Respiratory depression was defined as respiratory rate less than 10 times/min or the oxygen saturation decrease more than 5% compared with the baseline value.
Injection pain | From the injection of propofol/ciprofol to the end of the surgery, an average of 1 hour.
  Pain during injection of propofol/ciprofol

CONTACTS AND LOCATIONS:
Overall Officials: Jiangling Wang, Dr., Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Study protocol will be shared when asked